CLINICAL TRIAL: NCT05993611
Title: A First-in-Human Study to Evaluate the Safety, Feasibility and Tolerability of Allogeneic CD6 Chimeric Antigen Receptor T Regulatory Cells (CD6-CAR Tregs) in Patients With Chronic Graft-Versus-Host Disease (cGVHD) After Allogeneic Hematopoietic Cell Transplantation (alloHCT)
Brief Title: Allogeneic CD6 Chimeric Antigen Receptor T Regulatory Cells (CD6-CAR Tregs) for the Treatment of Patients With Chronic Graft Versus Host Disease After Allogeneic Hematopoietic Cell Transplantation
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: pending funding
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22375; NCI-2023-04067 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22375 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Chronic Graft Versus Host Disease; Hematologic and Lymphocytic Disorder; Steroid Refractory Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Hematologic Diseases | interventions — Biopsy; Specimen Handling; Immunotherapy, Adoptive; Leukapheresis; Spinal Puncture; Magnetic Resonance Spectroscopy; tafasitamab; Immunoglobulins; Disulfides; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CD6-CAR Treg, tafasitamab) (Experimental): Donors undergo leukapheresis over 2-4 hours for collection of PBMSc and the manufacturing of CD6-CAR Treg cells over 2 weeks. Patients then receive CD6-CAR Treg intravenously on day 0. Patients may also receive ablation tafasitamab IV post Treg cell infusion on days 1, 4, 8, 15, 22 for 1 cycle. If ablation is not complete by day 28, patients may receive an additional 1-2 cycles per investigator's discretion. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO, CT, and x-ray imaging during screening and as clinically indicated. Patients undergo blood specimen collection on study and during follow-up. Patients may undergo a biopsy on study as well as a lumbar puncture and MRI/CT as clinically indicated on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Biological: Chimeric Antigen Receptor T-Cell Therapy; Procedure: Computed Tomography; Procedure: Echocardiography; Other: Electronic Health Record Review; Procedure: Leukapheresis; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Biological: Tafasitamab; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Chimeric Antigen Receptor T-Cell Therapy — Given CD6-CAR Tregs IV
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell Therapy; Chimeric Antigen Receptor T-cell Infusion
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Other: Electronic Health Record Review — Ancillary studies
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI/CT
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Tafasitamab — Given IV
  Other Names: Immunoglobulin, Anti-(Human Cd19 Antigen) (Human-mus musculus Monoclonal MOR00208 Heavy Chain), Disulfide with Human-mus musculus Monoclonal MOR00208 .Kappa.-chain, Dimer; Monjuvi; MOR-00208; MOR00208; MOR208; Tafasitamab-cxix; XmAb5574
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of allogeneic CD6 chimeric antigen receptor T regulatory cells (CD6-CAR Tregs) in treating patients who have chronic graft versus host disease (cGVHD) after an allogeneic hematopoietic cell transplantation (HCT). An allogeneic HCT is an established treatment for benign or malignant blood and marrow conditions where healthy stem cells from a donor are infused into a patient to help the patient's bone marrow make more healthy cells and platelets. GVHD is a systemic disorder that occurs when the graft's immune cells recognize the host as foreign and attack the recipient's body cells. "Graft" refers to transplanted, or donated tissues, and "host" refers to the tissues of the recipient. It is a common complication after allogeneic HCT. The onset of cGVHD is usually within three years of transplantation and has some features of autoimmune diseases. A strategy that minimizes the incidence and severity of cGVHD, without other adverse effects, is needed to improve survival after allogeneic HCT. T regulatory cells are critical for controlling autoimmunity and maintaining immune homeostasis. Patients with active cGVHD have reduced numbers of T regulatory cells compared to patients without GVHD, suggesting that restoration of T regulatory cells in patients with active cGCHD is impaired and insufficient numbers may contribute to cGVHD. Therefore, therapies that augment numbers and function of T regulatory cells may promote tolerance and control of cGVHD. CAR T-cell therapy is a type of treatment in which T cells (a type of immune system cell) are taken from the blood and changed in the laboratory. The gene for a special receptor that binds to a certain protein, CD6, on the patient's cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion. CD6-CAR Tregs combines the CD6-targeted anti-inflammatory response with the immune regulatory properties of T regulatory cells which could generate a more potent and stable T regulatory cell population to promote immune tolerance and long-term disease control in cGVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if CD6-CAR Tregs administration is safe and tolerable in patients who developed chronic graft-versus-host disease (cGVHD), by evaluation of toxicities, including: type, frequency, severity, attribution, time course and duration.

II. To evaluate the feasibility to produce donor derived CD6-CAR Tregs.

SECONDARY OBJECTIVES:

I. Obtain preliminary evidence of CD6-CAR Tregs activity against cGVHD by estimating the response rate (as defined by 2014 National Institute of Health [NIH] consensus development project on clinical trials in cGVHD).

II. Evaluate changes in cGVHD severity using physician -reported cGVHD activity assessment form.

III. Evaluate changes in symptom activity using cGVHD activity assessment patient self-report.

IV. Evaluate failure-free survival (FFS). V. Quantify CD6-CAR Treg cells in peripheral blood. VI. Characterize and assess changes in immune biomarkers over time in blood samples.

EXPLORATORY OBJECTIVES:

I. Percent and counts from peripheral blood T cell subsets in hematopoietic stem/progenitor cell compartments to assess ability of CD6-CAR Tregs to suppress pathogenic T cell activity and proliferation.

II. Profile cytokine levels over time and changes to assess the ability of CD6-CAR Tregs to down-regulate proinflammatory cytokine production (IFNgamma, IL-6, TNFalpha) and adhesion molecules that promote pathogenic T cell.

III. For subjects who receive tafasitamab-cxix for CAR Treg ablation, describe the activity of infusional tafasitamab-cxix to eliminate transferred CD6 CAR Treg cells.

OUTLINE: This is a dose-escalation study of CD6-CAR Treg cells followed by a dose-expansion study.

Donors undergo leukapheresis over 2-4 hours for collection of peripheral blood mononuclear cells (PBMSc) and the manufacturing of CD6-CAR Treg cells over 2 weeks. Patients then receive CD6-CAR Treg intravenously on day 0. Patients may also receive ablation tafasitamab IV post Treg cell infusion on days 1, 4, 8, 15, 22 for 1 cycle. If ablation is not complete by day 28, patients may receive an additional 1-2 cycles per investigator's discretion. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO), computed tomography (CT), and x-ray imaging during screening and as clinically indicated. Patients undergo blood specimen collection on study and during follow-up. Patients may undergo a biopsy on study as well as a lumbar puncture and magnetic resonance imaging (MRI)/CT as clinically indicated on study.

After completion of study treatment, patients are followed up to 28 days, monthly for 1 year, and then yearly for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT (RECIPIENT) INCLUSION CRITERIA:
* All participants must have the ability to understand and the willingness to sign a written informed consent
* Participants must agree to allow the use of archival tissue from diagnostic biopsies.

  * If unavailable, exceptions may be granted with study PI approval Note: For research participants who do not speak English, a short form consent may be used with a City of Hope (COH) certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated full consent is processed
* Age >= 18 years
* Karnofsky performance status of >= 70%
* Received allogeneic hematopoietic stem cell transplantation (alloHCT) from matched related or haploidentical donor as part of treatment of hematologic disorders Note: The donor needs to consent for leukapheresis
* Clinical diagnosis of steroid-dependent or refractory, moderate to severe cGVHD

  * Steroid refractory cGVHD defined as having persistent signs and symptoms of cGVHD per institutional policy despite the use of prednisone for 2 months without complete resolution of signs and symptoms
* Estimated life expectancy > 90 days
* Stable dose of corticosteroids for >= 14 days prior to enrollment not exceeding 15mg/day of prednisone or equivalent + with up to 7ng/mL/day sirolimus with therapeutic drug monitoring
* Exposure to at least 1 of the Food and Drug Administration (FDA) approved tyrosine kinase inhibitor (TKI) therapies for cGVHD
* Naive to anti-CD6 therapy post most recent alloHCT
* Absolute neutrophil count (ANC) >= 1,000/mm^3 (without myeloid growth factors within 1 week of study entry) (performed within 28 days prior to enrollment)
* Platelets >= 50,000/mm^3 (performed within 28 days prior to enrollment) NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment
* Total bilirubin =< 2 mg/dL (exception permitted in patients with Gilbert's syndrome), unless hepatic dysfunction is a manifestation of presumed cGVHD) (performed within 28 days prior to enrollment) NOTE: Abnormal liver function tests (LFTs) (liver function panel) in the context of active cGVHD involving other organ systems may also be permitted if the treating physician documents the abnormal LFTs as being consistent with hepatic cGVHD and a liver biopsy will not be mandated in this situation
* Aspartate aminotransferase (AST) =< 3.0 x upper limit of normal (ULN) (performed within 28 days prior to enrollment)
* Alanine aminotransferase (ALT) =< 3.0 x ULN (performed within 28 days prior to enrollment)
* Creatinine clearance of >= 30 mL/min per 24-hour urine test or the Cockcroft-Gault formula (performed within 28 days prior to enrollment)
* Seronegative for human immunodeficiency virus (HIV) antigen/antibody (Ag/Ab) combo, hepatitis C virus (HCV)*, active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR]) (performed within 28 days prior to enrollment)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed OR
  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable
* Subjects must have negative QuantiFERON-tuberculosis (TB) Gold (QFTG) test (performed within 28 days prior to enrollment). Patients with positive QFTG test need clearance from infectious disease (ID) before enrollment
* Negative for coronavirus disease 2019 (COVID-19) within 72 hours of day 0 of protocol therapy (performed within 28 days prior to enrollment)
* Meets other institutional and federal requirements for infectious disease titer requirements Note Infectious disease testing to be performed within 28 days prior to start of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (performed within 28 days prior to enrollment) Note: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Cardiac function (12 lead-electrocardiography [ECG]): corrected QT interval (QTc) must be =< 480 msec (performed within 28 days prior to enrollment)
* Left ventricular ejection fraction > 40% (performed within 28 days prior to enrollment)
* Oxygen saturation 92% or above at room air or carbon monoxide diffusing capability test (DLCO) of 40% of best predicted (performed within 28 days prior to enrollment) Note: The above criteria only applies to participants who are not experiencing lung GVHD bronchiolitis obliterans syndrome (BOS)
* Agreement by females and males of childbearing potential* to use an effective method of birth control** or abstinence from sexual activity for the course of the study through at least 6 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

    * Effective birth control defined as hormonal and/or barrier contraception)
* ALLOGENEIC DONOR CRITERIA FOR APHERESIS DONATION:
* The identified donor must be the original donor whose stem cells were used for the research participant's alloSCT
* Karnofsky Performance Status (KPS) >= 70
* Age: >= 18 years
* The donor is approved and has completed the donor evaluation per institutional guidelines (as indicated in DACT 122 - Administrative Protocol for Allogeneic Hematopoietic Progenitor Cell, Apheresis [HPC(A)] Collections). Additionally, donor will also be screened for the following infectious diseases:

  * Epstein-Barr virus (EBV),
  * Human herpes virus 6, 7, and 8 (HHV6, HHV7, HHV8)
  * Parvovirus B19 Note: ID test results for EBV, HHV6, HHV7, HHV8 and Parvovirus B19 are not necessary to proceed with the apheresis procedure but do have to be resulted and negative before participant CAR Treg infusion

Exclusion Criteria:

* PATIENT (RECIPIENT) EXCLUSION CRITERIA:
* Immunosuppressive therapy within 28 days prior to enrollment (exception: corticosteroid)
* Concurrent other investigational agents, including biologics
* Vaccines within 28 days prior to enrollment
* Donor lymphocyte infusion within 100 days of enrollment
* No known contraindications to steroids or tocilizumab
* No current active malignancy* (Exception: Basal or squamous cell carcinoma)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Active uncontrolled infection requiring systemic antibiotics and/or anti-virals
* Other autoimmune/inflammatory disorders
* Clinically significant uncontrolled illness
* History of vascular disease (e.g., deep vein thrombosis, stroke)
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Uncontrolled atrial fibrillation or hypertension
* Females only: Pregnant or breastfeeding
* Inability to comply with protocol therapy and follow up visits
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-05-21 (Estimated); Study Completion 2028-05-21 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | From infusion of Allogeneic CD6 chimeric antigen receptor T regulatory cells (CD6-CAR Tregs) to day +28
  Toxicity will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0; cytokine release syndrome and immune effector cell associated neurotoxicity syndrome will be assessed per American Society for Transplantation and Cellular Therapy consensus criteria. Observed toxicities will be summarized by type, severity, date of onset, duration, reversibility, and attribution.
Feasibility as the ability to met at least 80% of the required cell dose at the assigned dose level | From infusion of CD6-CAR Tregs to day +28
  Will be estimated with 90% confidence interval (CI) overall and by dose level.
Feasibility as the ability to meet the required produce release criteria | From infusion of CD6-CAR Tregs to day +28
  Will be estimated with 90% CI overall and by dose level.

SECONDARY OUTCOMES:
CD6-CAR Treg activity | Up to 15 years
  As measured by changes in chronic graft versus host disease (cGVHD) severity.
Changes in cGVHD severity | Baseline up to 15 years
  Will be evaluated using cGVHD activity assessment patient self-report. Various graphical methods will be used to explore the association between immune response measures (at different time points and the changes over time) with changes in cGVHD severity.
Failure-free survival (FFS) | From infusion of CD6-CAR Tregs to start of new treatment for cGVHD, recurrence of malignancy, or death, whichever comes first, assessed at week 12 and 1-year follow-up
  Kaplan-Meier curve will be used to estimate FFS.
Relapse-free survival | From the start of treatment to the date of death, disease relapse, or last follow-up whichever occurs first, assessed up to 15 years
CD6-CAR Treg persistence | Up to 15 years
  Immunophenotyping (CD19t, CD3, CD4, CD8) (fluorescence-activated cell sorting/ co-detection by indexing), cytokine release syndrome (including TNF-alpha, IL-2, IL-6, IL-10 and IFN-gamma) (multiplex assay), immunogenicity (anti-CAR antibodies) (enzyme-linked immunosorbent assay)
Changes in immune biomarkers over time | Baseline up to 15 years
  Descriptive statistics and graphics will be used to characterize and plot the specific time trend for each marker of the immune response. Various graphical methods will be used to explore the association between these immune response measures (at different time points and the changes over time) with changes in cGVHD severity.
Infectious complications | From day 1 to day 28 of CD6-CAR Treg infusion, up to 15 years
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any. This data will be captured via case report form and will be collected from day 1 to day 28 of alloCD6-CAR Treg infusion and will follow the same data collection intervals as the toxicity and adverse event data. Severity of the infections will be graded by CTCAE v5.0 and Blood and Marrow Clinical Trials Network.

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Salhotra, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States